CLINICAL TRIAL: NCT06872502
Title: Mindfulness-based Intervention for Psychophysical Well-Being in the Italian Elderly
Brief Title: Meditation and Psychophysical Well-Being in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Teresa Fazia, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1Med_b
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Loneliness; Psychophysical Well-being
Keywords: mindfulness; elderly; loneliness; social isolation; wellbeing
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: The study involves two groups: one receiving the mindfulness-based intervention and a control group (waiting-list control).
  Participants are randomized into these two groups and followed in parallel without switching between conditions.
  The outcomes are measured before and after the intervention, comparing the effects between the two groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Outcomes Assessor and Data Analyst are blinded to group allocation. The meditation trainer is aware of the group assignment but does not have access to the outcome measures. participants are not blinded to their assigned group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention Group (Experimental): Participants in this group will undergo a mindfulness-based meditation intervention called Integral Meditation (IM). The intervention consists of 12 in-person sessions over six weeks, with each session lasting one hour, twice per week. The meditation techniques will include focused breathing, body relaxation, emotional awareness, and acceptance exercises.
  Interventions: Behavioral: Mindfulness-Based Meditation (Integral Meditation - IM)
- Waiting-List Control Group (No Intervention): Participants in this group will not receive any intervention during the study period. They will be placed on a waiting list and instructed to refrain from any meditation or mindfulness-based activities until the study is completed. This group serves as a passive control to evaluate the effectiveness of the mindfulness-based intervention by comparing pre- and post-intervention measures.

INTERVENTIONS:
Behavioral: Mindfulness-Based Meditation (Integral Meditation - IM) — The intervention consists of 12 in-person mindfulness-based meditation sessions over a period of six weeks, with each session lasting one hour, twice per week. The practice, called Integral Meditation (IM), includes focused breathing, body relaxation, emotional awareness, and acceptance exercises.
  Other Names: Integral Meditation (IM)
  Arms: Mindfulness-Based Intervention Group

SUMMARY:
The goal of this experimental study is to assess whether a mindfulness-based meditation intervention can reduce loneliness and improve psychophysical well-being in older adults (aged 65 and above).

The main questions it aims to answer are:

* Does the intervention reduce the perception of loneliness in older adults? (primary outcome)
* Does it improve various aspects of psychological well-being, including social isolation, depression, life satisfaction, mindfulness, emotional regulation, self-acceptance, and sleep quality? (secondary outcomes) Researchers will compare the intervention group with a passive control group (waiting-list control) to determine whether the mindfulness-based intervention leads to significant improvements in the measured outcomes.

Participants will:

Complete baseline assessments, including neuropsychological tests and validated questionnaires, before the intervention.

Undergo a 12-session mindfulness-based intervention over 6 weeks, consisting of guided breathing, focused attention, physical relaxation, and emotional awareness exercises.

Complete post-intervention assessments to measure changes in their psychological and physiological well-being.

DETAILED DESCRIPTION:
The aging of the population is now a global phenomenon, and according to the United Nations World Population Prospects 2024, it is estimated that the population over the age of 65 could reach ~24% by the end of this century. Italy ranks as the second country in the world with the highest proportion of elderly citizens. According to recent ISTAT data, individuals over 65 represent ~25% of the total population. This demographic imbalance, strongly skewed toward older age groups, reflects both a low birth rate and increased longevity.

Unfortunately, at least nine million elderly individuals in Italy live alone or are at risk of social isolation. According to data from the "Passi d'Argento" surveillance system of the Italian National Institute of Health (Istituto Superiore di Sanità), this phenomenon affects 1 in 7 people over 65. Social isolation significantly impacts healthy aging, compromising both physical and mental well-being.

Social isolation consists of two components: an objective one and a subjective one, namely loneliness. These two dimensions do not always correlate and affect health through different pathways: the former is more closely linked to physical health, while the latter is primarily associated with mental health.

Several risk factors contribute to this condition (e.g., educational level, environment in which a person was raised, comorbidities, income, etc.), also influencing coping mechanisms. Addressing this social and economic challenge requires timely and sustainable interventions. In this context, mindfulness represents a promising therapeutic and preventive tool.

Mindfulness-based interventions are easily accessible, simple to implement, and have a low economic impact, while promoting both physical and mental health. They foster psychological well-being and personal growth, encouraging a non-judgmental awareness of the present moment. Mindfulness can help older adults accept the changes and losses associated with aging, enhancing self-awareness and developing new coping strategies. Furthermore, mindfulness may serve as a tool to recognize and understand loneliness, potentially transforming it into an opportunity for personal growth.

By promoting active listening, empathy, and self-esteem, mindfulness can also contribute to improving the quality of social relationships. However, studies exploring the effects of mindfulness on loneliness-particularly in older adults-are still limited and often involve small sample sizes and lack comprehensive sociodemographic data.

The objective of this study is to evaluate the impact of a mindfulness-based meditation intervention on the sense of loneliness (primary outcome) as well as on various domains of psychophysical well-being in older adults.

Specifically, the following hypotheses will be tested:

i) The intervention reduces the sense of loneliness (primary outcome); ii) It decreases objective social isolation; iii) It lowers depression levels, contributing to an overall improvement in psychological well-being; iv) It enhances mental well-being and life satisfaction; v) It improves mindfulness and promotes emotional regulation; vi) It fosters greater self-acceptance in terms of body appreciation and enhances self-esteem; vii) It improves sleep quality.

The target population will consist of older adults aged 65 and above, recruited on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the Italian language
* Age ≥ 65 years
* No cognitive impairment, as measured by the Addenbrooke's Cognitive Examination (ACE-R)

Exclusion Criteria:

* Presence of severe mental disorders and/or significant medical conditions
* Substance dependence

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Perceived Loneliness | Baseline (T0), post-intervention (6 weeks, T1)
  The primary outcome is the change in perceived loneliness as measured by the UCLA Loneliness Scale (Version 3). Scores range from 20 to 80, with higher scores indicating greater loneliness. A significant reduction in scores post-intervention would suggest an improvement in loneliness perception.

SECONDARY OUTCOMES:
Reduction in Objective Social Isolation Reduction in Objective Social Isolation Reduction in Objective Social Isolation Reduction in Objective Social Isolation Reduction in Objective Social Isolation | Baseline (T0), post-intervention (6 weeks, T1)
  we will evaluated changes in social isolation assessed using the Lubben Social Network Scale (LSNS-6), which evaluates the size and frequency of participants' social networks. Higher scores indicate greater social connectivity.
Reduction in Depressive Symptoms | Baseline (T0), post-intervention (6 weeks, T1)
  we will evaluate changes in depression levels assessed using the Geriatric Depression Scale (GDS-15). Higher scores indicate greater depressive symptoms, while a reduction in scores suggests improved mental well-being.
Improvement in Well-being and Life Satisfaction | Baseline (T0), post-intervention (6 weeks, T1)
  We will evaluate subjective well-being and life satisfaction using the Satisfaction with Life Scale (SWLS) questionnaire and the Warwick-Edinburgh Mental Well-Being Scale(WEWBS). Higher scores indicate greater satisfaction with life.
Increase in Mindfulness and Emotional Regulation | Baseline (T0), post-intervention (6 weeks, T1)
  We will evaluate mindfulness levels using the Five Facet Mindfulness Questionnaire (FFMQ) and emotional regulation using the Emotion Regulation Questionnaire (ERQ). Higher scores indicate improved mindfulness and emotion regulation
Improvement in Self-Esteem and body appreciation | Baseline (T0), post-intervention (6 weeks, T1)
  We will evaluate Self-esteem via the Rosenberg Self-Esteem Scale (RSES) and via the Body Appreciation Scale we will assess the level of appreciation towards one's own body. Higher scores indicate greater self-esteem and body appreciation.
Improvement in Sleep Quality | Baseline (T0), post-intervention (6 weeks, T1)
  Using the Pittsburgh Sleep Quality Index (PSQI), we will evaluate subjective sleep quality. Higher scores indicate worse sleep quality, while a reduction in scores suggests improved sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavia, Pavia, Italy